CLINICAL TRIAL: NCT04248790
Title: Design and Development of a Mobile App to Improve Adherence to Pre-exposure Prophylaxis in Men Who Have Sex With Men: A Pilot Study
Brief Title: Design and Development of a Mobile App to Improve Adherence to Pre-exposure Prophylaxis in Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng Kung University (Other)
Collaborators: National Cheng-Kung University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); National Tsing Hua University (Other)
Responsible Party: Principal Investigator, Carol Strong, Associate Professor, National Cheng Kung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TaiwanUPrEPU; MOST 108-2636-B-006-004 (Other Grant/Funding Number: Taiwan Ministry of Science and Technology)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections; Pre-Exposure Prophylaxis
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: the mobile App (Experimental): Participants in the intervention arm will receive access to all the app capabilities. The app features include information on HIV testing locations, sex and PrEP diary and reminder of taking PrEP.
  Interventions: Behavioral: mobile app to improve adherence to PrEP self-management

INTERVENTIONS:
Behavioral: mobile app to improve adherence to PrEP self-management — Access to the mobile app which includes the sex and PrEP diary, information on HIV/STI testing, PrEP reminders and geo-location features.

SUMMARY:
This study is testing feasibility and acceptability of a theoretically based mobile application (app), UPrEPU, to increase adherence to pre-exposure prophylaxis (PrEP) among men who have sex with men (MSM) to prevent human immunodeficiency virus (HIV).

DETAILED DESCRIPTION:
This study aims to develop an effective mobile application (app), UPrEPU to recognize the factors and decisions that affect PrEP adherence in high-risk populations to improve PrEP adherence. Key components of the app include a sex/PrEP diary using ecological momentary assessment to facilitate accurate data collection; PrEP taking reminder; HIV and sexually transmitted infections (STI) testing information and reminders; HIV and PrEP information and videos; geo-location.

After eligible PrEP candidates agree to participate in the study, we will ask participants to install the app. Then, we will begin to collect their sexual diary and PrEP taking log via ecological momentary assessment. Participants will also complete monthly assessments. The monthly follow-up will test HIV/STI and drug concentration. The participants will be interviewed for difficulties when they use our app and giving feedback on it.

ELIGIBILITY:
Inclusion criteria:

* Male.
* Aged 20 or above.
* Resides in Taiwan and able to understand, read, and speak Mandarin Chinese.
* Remains HIV negative prior to and during the study period.
* The results of the laboratory tests are eligible to initiate PrEP.
* Currently taking PrEP or willing to initiate PrEP.
* Reports having 4 times or above anal sex with men in the past month.
* Owns an Android or Apple operating system (iOS) smartphone and willing to download the study app.
* Willing to wear the device we provided during the study period.

Exclusion criteria:

* With abnormal kidney function (creatinine clearance rate ≦ 60 mL/minute).
* Currently on medication that might interact with PrEP, such as drugs contain lamivudine in the pre-PrEP assessment.

Ages: 20 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Usability | 4 months
  Scores on system usability scale (SUS) for this app at the first month and the fourth month.
Feasibility: data based on the app analytics | 4 months
  1. Frequency of app log-in;
  2. Use of app components such as PrEP-taking and sex behavior reports;
  3. Duration of app use
Efficacy of adherence monitoring | 4 months
  Measuring the Tenofovir (TDF) and Emtricitabine (FTC) drug concentration in dried blood spot (DBS) samples to compare with self-report data

SECONDARY OUTCOMES:
Feasibility: data from qualitative interviews | 4 months
  1. any technical challenges participants may have encountered;
  2. recommendations for the app improvement;
  3. users' satisfaction and comfort in using this app

CONTACTS AND LOCATIONS:
Overall Officials: Carol Strong, PhD, Principal Investigator — National Cheng Kung University
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan, Tainan
  - Taipei city hospital (Renai Branch), Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strong C, Wu HJ, Tseng YC, Yuan CW, Yu YF, Liao JC, Chen YW, Hung YC, Li CW, Huang PH, Ko NY, Ku SW. Mobile App (UPrEPU) to Monitor Adherence to Pre-exposure Prophylaxis in Men Who Have Sex With Men: Protocol for a User-Centered Approach to Mobile App Design and Development. JMIR Res Protoc. 2020 Dec 1;9(12):e20360. doi: 10.2196/20360. PMID 33258793

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04248790/Prot_SAP_000.pdf